CLINICAL TRIAL: NCT03501511
Title: Comparison of Two Health Education Modalities for Safe Ramadan Fasting in People With Type 1 Diabetes
Brief Title: Health Education During Ramadan Fasting in Type 1 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Dr.Yara Eid, Professor of Internal Medicine-Endocrinology and Metabolism Unit , Ain-Shams University, Ain Shams University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: FMASU/MS 20/2017
Record Dates: First submitted 2018-04-10; First posted 2018-04-18 (Actual); Last update posted 2018-06-29 (Actual); Status verified 2018-06

CONDITIONS: Diabetes Mellitus, Type 1; Fasting
Keywords: Diabetes MellitusType1;Fasting;Health Education;Hypoglycemia
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Fasting

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IDF modules (Active Comparator): Diabetes educations using IDF Arabic translated modules
  Interventions: Behavioral: IDF modules
- Conversational Maps (Experimental): Diabetes Educations using Ramadan fasting conversational maps (Arabic maps)
  Interventions: Behavioral: Conversational Maps

INTERVENTIONS:
Behavioral: IDF modules — Patients in this arm will receive Pre-Ramadan education using IDF module for 4 weeks prior to Ramadan fasting
  Arms: IDF modules
Behavioral: Conversational Maps — Patients in this arm will receive Pre-Ramadan Education using Ramadan Fasting Diabetes conversation map for 4 weeks prior to Ramadan fasting
  Arms: Conversational Maps

SUMMARY:
Adult Muslims are obliged to start fasting during the month of Ramadan. Fasting entails refraining from all food, drink, tablets and injections(vitamins & fluids) between sunrise and sunset; a period which varies by geographical location and season.

People with type 1 Diabetes are among those who are risky to fast this holy month in the Muslim faith and thus are exempted from fasting. Yet many patients fast in spite of medical advice and religious exemption and for those patients, healthcare professionals should provide the utmost care and continuous diabetes education.

Different diabetes education modalities exist like DSME (Diabetes self-management education with proven efficacy. One modality is the Diabetes Conversation Map which delivers diabetes education interactively through a series of maps that address different issues in diabetes management and includes a specially designed Ramadan map.

In this study, two modalities of Diabetes focused Ramadan education will be compared regarding aiding patients to fast Ramadan safely. One modality will be Diabetes conversation maps and the other the International Diabetes Federation Education modules.

DETAILED DESCRIPTION:
Adult Muslims are obliged to start fasting during the month of Ramadan. Fasting entails refraining from all food, drink, tablets and injections(vitamins & fluids) between sunrise and sunset; a period which varies by geographical location and season. Although exempt, many diabetics refuse to take this concession as they feel psychologically & spiritually inclined to fast along with other Muslims.

Fasting at Ramadan carries a very high risk for people with T1DM. This risk is particularly exacerbated in poorly controlled patients and those with limited access to medical care, hypoglycemic unawareness, unstable glycemic control, or recurrent hospitalizations.

Structured education interventions have been endorsed by the National Institute for Health and Clinical Excellence as important in empowering patients to improve their jour¬ney with diabetes. In a large observational study, patients who fasted during Ramadan without attending a structured education session had a fourfold increase in hypoglycae¬mic events, whereas those who attended an education pro¬gramme focusing on Ramadan had a significant decrease in hypoglycemic events.

Conversation Map aims to help people with diabetes experience a healthier Ramadan. The interactive Map covers a number of topics including understanding the risks and complications of fasting and the importance of creating a diabetes management plan during this time.

ELIGIBILITY:
Inclusion Criteria:

1. Patients are intending to fast .
2. Duration of diabetes is more than 5 years .
3. Insulin regimen is basal-bolus .

Exclusion Criteria:

1. Acute complications as major events of hypoglycemia or DKA during the last 3 months before Ramadan .
2. Pregnancy .
3. Previous stroke, MI, or unstable angina .

Ages: 16 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 53 (Actual)
Dates: Start 2018-04-07 (Actual); Primary Completion 2018-06-28 (Actual); Study Completion 2018-06-28 (Actual)

PRIMARY OUTCOMES:
Hypoglycemia | Detected through Self monitoring of blood glucose during 4 weeks of Ramadan fasting
  Rate of attacks of hypoglycemia during Ramadan

SECONDARY OUTCOMES:
Insulin Dose Adjustment | During 4 weeks of Ramadan fasting
  percent reduction or increase in basal and bolus insulin dose during month of Ramadan
Body Weight Change | Measurement of body weight prior month of Ramadan and after the month of Ramadan
  Increase or decrease of body weight at the end of Ramadan month fasting
Number of successful fasting days | During 4 weeks of Ramadan fasting
  Number of days completed fasting per patient

CONTACTS AND LOCATIONS:
Overall Officials: Yara M Eid, MD, Principal Investigator — Ain-Shams University -Faculty of Medicine; Manal A AbuShady, MD, Study Chair — Ain-Shams University -Faculty of Medicine; Mona M AbdelSalam, MD, Study Director — Ain-Shams University -Faculty of Medicine
Locations (1):
- Ain-Shams University-Faculty of Medicine- Ain-Shams University Hospitals -Internal Medicine Department -Endocrinology and Metabolism Unit, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided